CLINICAL TRIAL: NCT04058210
Title: VX-445/TEZ/IVA Triple Combination Expanded Access Program for Patients 12 Years of Age and Older With Cystic Fibrosis Who Are Heterozygous for F508del and a Minimal Function CFTR Mutation
Brief Title: VX-445/TEZ/IVA Expanded Access Program for Cystic Fibrosis (CF) Patients Heterozygous for F508del Mutation and a Minimal Function Mutation (F/MF Genotypes)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: VX18-445-901
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination tablet for oral administration.
  Other Names: elexacaftor/tezacaftor/ivacaftor; VX-445/VX-661/VX-770
Drug: IVA — 150-mg tablet for oral administration.
  Other Names: ivacaftor; VX-770

SUMMARY:
The purpose of this program is to provide elexacaftor(ELX, VX-445)/tezacaftor(TEZ)/ivacaftor(IVA) combination therapy to CF patients in critical need who are 12 years of age and older, heterozygous for F508del and a minimal function (MF) mutation in response to unsolicited physician requests.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have F/MF genotypes AND who meet at least 1 of the following criteria:

* The percent predicted forced expiratory volume in 1 second (ppFEV1) is <40 for a minimum of 2 months before the date of the request, OR
* Documentation of being active on a lung transplant waiting list or documentation of being evaluated for lung transplantation, but deemed unsuitable because of contraindications

Exclusion Criteria:

1. Patients with severe hepatic impairment (Child-Pugh Class C)
2. History of any other comorbidity that, in the opinion of the treating physician, might pose undue risk in administering ELX/TEZ/IVA to the patient
3. Pregnancy

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult